CLINICAL TRIAL: NCT03573466
Title: Presymptomatic Neuromuscular Junction Defects and Compensatory Mechanisms in Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Presymptomatic Neuromuscular Junction Defects and Compensatory Mechanisms in ALS
Acronym: PRE-ALS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P171004J; 2018-A00573-52 (Other: ANSM)
Record Dates: First submitted 2018-06-15; First posted 2018-06-29 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Motor Neuron; Neuromuscular Junction
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amyotrophic Lateral Sclerosis (Experimental)
  Interventions: Procedure: Muscle biopsy

INTERVENTIONS:
Procedure: Muscle biopsy — A motor point biopsy of deltoid muscle will be carried out at the time of inclusion using a standardized procedure, as routinely performed. Muscle samples will be removed from the deltoid muscle by open biopsy under local anaesthesia. The region containing NMJs will be determined by the small twitch provoked by the tip of the scalpel on the surface of the muscle fascicles.

SUMMARY:
Denervation of neuromuscular junctions (NMJs) and initial compensatory reinnervation is the earliest pathological event in various motor neuron disease models, occurring far before motor symptom onset. In patients harboring genetic mutations responsible for Amyotrophic Lateral Sclerosis (ALS), identification of early, pre-symptomatic, NMJ pathological events and compensatory mechanisms could lead to the development of new treatments to prevent motor functional impairment.

The aims of our study are thus:

1. To investigate and characterize early, presymptomatic, defects of NMJ morphology in pre-manifest C9ORF72 or SOD1 mutation carriers;
2. To investigate and quantify reinnervation at the level of NMJs in these subjects;
3. To identify muscle molecular dysregulated pathways involved in the development of NMJ alterations and the development / maintenance of compensatory collateral reinnervation.

DETAILED DESCRIPTION:
The neuromuscular junction (NMJ), where the axon terminal connects the motor endplate of the muscle fiber, is the first structure affected in various Amyotrophic Lateral Sclerosis (ALS) rodent models. In these models, NMJ denervation and initial compensatory reinnervation are the earliest pathological event. These NMJ morphological defects occur far before changes can be seen at the level of motor neuron cell bodies and motor symptom onset. In these rodent models, there is thus a "latency phase" of the disease.

In ALS patients, the onset of symptoms is believed to occur when approximately 50 to 80% of motor neurons are lost and it has been suggested that the disease may have a prolonged preclinical period. After clinical onset of the disease, the existence of striking NMJ morphological defects and compensatory reinnervation of endplates has been shown in muscle of ALS patients, but their occurrence at the presymptomatic stage has never been investigated. As in animal models, at the subclinical onset of the disease, efficient reinnervation of NMJs could compensate for the loss of motor neurons and subjects would remain free of any motor symptom. As the destruction of NMJs progresses, compensation would become ineffective, leading to progressive muscle weakness and clinical onset of the disease. Identification of early, pre-symptomatic, NMJ pathological events and compensatory mechanisms could thus lead to the development of new treatment strategies to prevent motor functional impairment.

In human, the "latency phase" of the disease can be investigated in pre-manifest ALS mutation carriers. Indeed, in a population of asymptomatic carriers of C9ORF72 or SOD1 mutations (two of the main genes associated with familial ALS), a dysregulation of circulating microRNAs has been found long before the estimated time window of disease symptom onset.

The objectives of the PRE-ALS study are:

Primary objective: to investigate and characterize early, preclinical defects of NMJ morphology in muscle specimens from pre-manifest C9ORF72 or SOD1 mutation carriers;

Secondary objectives:

* to investigate and quantify reinnervation at the level of NMJs in these subjects; and
* to identify muscle dysregulated pathways involved in the development of NMJ alterations and the development / maintenance of compensatory collateral reinnervation.

For this purpose, ten subjects with mutations in one of two major ALS-associated genes - C9ORF72 and SOD1- free from any motor symptom, will be included in the study. These subjects, diagnosed on the basis of presymptomatic DNA tests performed in the context of familial ALS or familial frontotemporal dementia linked to C9ORF72 expansion (C9-FTD), will be recruited from the Paris ALS center (Dr Salachas) and the Reference Centre for Rare Dementias (Dr Le Ber). Subjects harboring mutations in the C9ORF72 gene with only moderate cognitive impairment may also be included if they are free of motor involvement after neurological examination.

Subjects will be clinically and neurophysiologically followed-up during 18 months after inclusion in the study:

* Muscle strength will be measured by manual muscle testing according to the grading system of the Medical Research Council;
* Functional motor impairment will be assessed using the widely used revised ALS Functional Rating Scale (ALSFRS-R), a 12-item scale that rates the performance of activities of daily living;
* Motor neuron loss will be evaluated using Motor Unit Number Index (MUNIX), a validated method to assess number and size of motor units in ALS patients.

A muscle biopsy will be performed to investigate potential morphological defects at the level of NMJs. The morphology of NMJs will be analyzed using confocal microscopy after immunostaining and collateral reinnervation will be quantified for each subject. Dysregulated intracellular signaling pathways potentially implicated in preclinical structural defects of NMJs and / or reinnervation will be investigated in parallel.

To date, the PRE-ALS study will be the first to investigate preclinical changes of NMJs in presymptomatic ALS mutation carriers and to identify muscle compensatory mechanisms allowing preservation of motor function. This work should pave the way to identification of new therapeutic strategies in order to prevent the occurrence of strength loss in ALS mutations carriers and limit muscle wasting in sporadic ALS patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects harboring a mutation in C9ORF72 or SOD1 gene
* Without any functional motor complaint and clinical motor deficit at neurological examination
* Aged 30 to 70 (inclusive).
* Patients covered by the social insurance system

Exclusion criteria:

* Any motor deficit
* Any significant cognitive or psychiatric impairment leading to limitation in decision making capacity
* Inability to give informed consent
* Patient unable to contact or to be contacted by the investigator in case of emergency
* Women who are pregnant or nursing, or without effective contraceptive method
* Concomitant medication contraindicating muscle biopsy (platelet suppressive agents, oral anticoagulant therapy)
* Medical condition contraindicating muscle biopsy (hypocoagulative disease, allergy to anaesthetic drugs, acute intermittent porphyria)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2023-05-25 (Estimated); Study Completion 2023-05-25 (Estimated)

PRIMARY OUTCOMES:
Quantification of neuromuscular junctions innervation | 18 month
  Quantification of innervation by confocal microscopy will be performed by classifying neuromuscular junctions observed in each biopsy specimen according to the relationship between the intrasynaptic axonal branches and the postsynaptic membrane in four categories: "normal", "denervated", "partially innervated", or "reinnervated"

CONTACTS AND LOCATIONS:
Overall Officials: Gaelle BRUNETEAU, BRUNETEAU, Principal Investigator — APHP
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No